CLINICAL TRIAL: NCT03024125
Title: Effect of Normal and High Protein Diets in Lean Mass, Adiposity, and Strength in Postmenopausal Women Practitioners of Resistance Exercise
Brief Title: High vs Normal Protein Diets, Resistance Exercise, Lean Mass and Strength Gains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Erick Prado de Oliveira, PhD, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.733.512
Record Dates: First submitted 2016-10-31; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Sarcopenia
Keywords: lean mass; postmenopausal; protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High protein diet (HP) (Experimental): Diet with 1.2 protein g/kg body mass/day for postmenopausal women practitioners of resistance exercise. The physical strength training will be performed equally by both groups
  Interventions: Other: High protein; Other: Training
- Normal protein diet (NP) (Placebo Comparator): Diet with 0.8 protein g/kg body mass/day for postmenopausal women practitioners of resistance exercise. The physical strength training will be performed equally by both groups
  Interventions: Other: Normal protein; Other: Training

INTERVENTIONS:
Other: High protein — To observe the effect of a high protein (HP) diet over muscle mass, fat mass, and strength changes, focusing in differences between the NP and HP groups.
  Arms: High protein diet (HP)
Other: Normal protein — To observe the effect of a normal protein (NP) diet over muscle mass, fat mass, and strength changes
  Arms: Normal protein diet (NP)
Other: Training — The physical strength training will be performed equally by both groups, containing exercises for upper and lower limbs and aiming for hypertrophy.

SUMMARY:
This study evaluates the effect of different types of diets (high and normal protein) on lean and fat mass, and strength in postmenopausal women practitioners of resistance exercise. Two groups will be created: high protein (1.2 protein g/body mass/day) and normal protein (0.8 protein g/body mass/day). The same training will be performed for both groups.

DETAILED DESCRIPTION:
Both groups will undergo the same training protocol, differing only on the protein content of the diet. The dietary assessment will be made through the 24-hour food recall, being conducted at the beginning, middle and end of the intervention. Resistance exercises for upper and lower limbs will be performed, at 70% of one repetition maximum. SPPB, tug, 6-minutes and 400 meters will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women in the postmenopausal period (menopausal for at least one year, confirmed by laboratory diagnostic tests menopause - LH and high FSH and estradiol decreased);
* Healthy;
* Who agree to participate and sign the consent term.

Exclusion Criteria:

* The one who does not provide the necessary information for the development of the study;
* Present orthopedic limitations;
* Patients with previously diagnosed and treatment of diseases such as type II diabetes mellitus, hypertension and cardiovascular disease.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Changes in the lean mass of postmenopausal women practicing strength exercise | Before and immediately after the intervention (initial moment and 10 weeks after start of the intervention)

SECONDARY OUTCOMES:
Changes in the fat mass of postmenopausal women practicing strength exercise | Before and immediately after the intervention (initial moment and 10 weeks after start of the intervention)
Changes on strength of postmenopausal women practicing strength exercise | Before and immediately after the intervention (initial moment and 10 weeks after start of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Erick P de Oliveira, PhD, Principal Investigator — Federal University of Uberlandia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nahas PC, Rossato LT, Martins FM, Souza AP, de Branco FMS, Carneiro MAS, Teixeira KRC, Orsatti FL, de Oliveira EP. Moderate Increase in Protein Intake Promotes a Small Additional Improvement in Functional Capacity, But Not in Muscle Strength and Lean Mass Quality, in Postmenopausal Women Following Resistance Exercise: A Randomized Clinical Trial. Nutrients. 2019 Jun 13;11(6):1323. doi: 10.3390/nu11061323. PMID 31200437
- [Derived] Rossato LT, Nahas PC, de Branco FMS, Martins FM, Souza AP, Carneiro MAS, Orsatti FL, de Oliveira EP. Higher Protein Intake Does Not Improve Lean Mass Gain When Compared with RDA Recommendation in Postmenopausal Women Following Resistance Exercise Protocol: A Randomized Clinical Trial. Nutrients. 2017 Sep 12;9(9):1007. doi: 10.3390/nu9091007. PMID 28895933